CLINICAL TRIAL: NCT01771172
Title: Acute Subcutaneous Defibrillation
Acronym: ASQ
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQ
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Ventricular Arrhythmias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the defibrillation efficacy of a subcutaneous defibrillation system.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing implant of a commercially approved ICD system
* Subject must be willing to provide Informed Consent
* Subject must be > 18 years old

Exclusion Criteria:

* Subject with impaired kidney function as measured by a glomerular filtration rate (eGFR) estimate < 29 mls/min/1.73m2 (recorded in the last six months)
* Subject has high risk of infection
* Subject has EF < 15%
* Subject at high risk of stroke
* having a device replacement
* Subject with an implanted active non-ICD device, cardiac or non-cardiac (e.g., Neuro stimulator, Pacemaker)
* Subject is indicated for CRT
* Subject is pacemaker dependent
* Subject enrolled in a concurrent study that may confound the results of this study
* Subject has medical conditions that would limit study participation
* Subject is pregnant
* Subject meets exclusion criteria required by local law (e.g. age, breast feeding, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects may be either male or female, and must meet all of the inclusion criteria and none of the exclusion criteria of the study
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Republican Scientific and Practical Center Cardiology, Minsk, Belarus
- Rigshospitalet, Copenhagen, Denmark
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- Slovak Medical University, Bratislava, Slovakia, Slovakia
- United Kingdom (3):
  - Dudley Group NHS-Russells Hall Hospital, Dudley
  - King's College Hospital, London
  - Southhampton General Hospital, Southhampton

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Defibrillation Testing
Started | 48
Completed | 46
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Acute Defibrillation Testing
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Subjects Will Demonstrate a Successful Defibrillation Outcome if They Have 2 Successful Defibrillation Shocks With the Research System.
Time Frame: within the first day
Measure: Number; unit: percentage of success
Arm/Group | Acute Defibrillation Testing
Number analyzed (Participants) | 35
percentage of success | 85.7

ADVERSE EVENTS:
Arm/Group | Acute Defibrillation Testing
Serious Adverse Events (participants affected / at risk) | 9/50
Other Adverse Events (participants affected / at risk) | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Defibrillation Testing (N=50)
Implant site infection (Skin and subcutaneous tissue disorders) | 2 (2)
Post Procedural Hematoma (Blood and lymphatic system disorders) | 2 (2)
Anaphylactic reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Adverse drug reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Defibrillation Testing (N=50)
Post Procedural Hematoma (Blood and lymphatic system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No